CLINICAL TRIAL: NCT05211128
Title: The Evolving Use of Robotic Surgery: A Population-based Analysis
Brief Title: The Evolving Use of Robotic Surgery
Status: Completed | Type: Observational
Sponsor: Sunnybrook Health Sciences Centre (Other)
Collaborators: University of Toronto (Other); Unity Health Toronto (Other); Western University (Other); McMaster University (Other); University of Ottawa (Other); Saskatchewan Cancer Agency (Unknown)
Responsible Party: Sponsor
Other Study IDs: 2019 0990 194 000
Record Dates: First submitted 2022-01-14; First posted 2022-01-27 (Actual); Last update posted 2022-01-27 (Actual); Status verified 2022-01

CONDITIONS: Surgery
Keywords: Robotic surgery
MeSH Terms: interventions — Robotic Surgical Procedures; Conversion to Open Surgery; Laparoscopy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Radical prostatectomies
  Interventions: Procedure: Robotic Surgery; Procedure: Open Surgery; Procedure: Laparoscopic Surgery
- Total hysterectomies
  Interventions: Procedure: Robotic Surgery; Procedure: Open Surgery; Procedure: Laparoscopic Surgery
- Thoracic lobectomies
  Interventions: Procedure: Robotic Surgery; Procedure: Open Surgery; Procedure: Laparoscopic Surgery
- Partial nephrectomies
  Interventions: Procedure: Robotic Surgery; Procedure: Open Surgery; Procedure: Laparoscopic Surgery

INTERVENTIONS:
Procedure: Robotic Surgery — Surgical procedure using robotic technologies.
Procedure: Open Surgery — Surgical procedure using a large, open cut in the skin.
Procedure: Laparoscopic Surgery — Surgical procedure using small incisions and trochars.

SUMMARY:
A retrospective, population-based analysis examining the rates of robotic surgery between the years of 2009 - 2018.

DETAILED DESCRIPTION:
A retrospective, population-based analysis examining the rates of robotic surgery in Ontario between the years of 2009 - 2018. The purposes of the study were (i) to describe temporal trends and (ii) patient- and system-level determinants of receiving robotic compared to open or laparoscopic surgery.

ELIGIBILITY:
Inclusion Criteria:

* Minimum 18 years old
* Received an elective radical prostatectomy, total hysterectomy, partial nephrectomy, or thoracic lobectomy using an open, laparoscopic or robotic approach between 2008-2018

Exclusion Criteria:

* Non-Ontario residents
* Non-elective procedure
* Patients without OHIP eligibility
* Patients who had an identical procedure in the previous two years

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Ontario adults that received an elective radical prostatectomy, total hysterectomy, partial nephrectomy, or thoracic lobectomy using an open, laparoscopic or robotic approach between 2008-2018.
Sampling Method: Non-Probability Sample
Enrollment: 123074 (Actual)
Dates: Start 2018-07-01 (Actual); Primary Completion 2021-06-01 (Actual); Study Completion 2021-06-01 (Actual)

PRIMARY OUTCOMES:
Temporal trends | 2009 - 2018
  To describe temporal trends in robotic surgery

OTHER OUTCOMES:
Determinants of surgery type | 2009 - 2018
  To identify patient- and system-level determinants of receiving robotic compared to open or laparoscopic surgery

CONTACTS AND LOCATIONS:
Locations (1):
- Sunnybrook Health Sciences Centre, Toronto, Ontario, Canada